CLINICAL TRIAL: NCT00980447
Title: A Multicenter, Non-Blinded, Dose Escalation Study to Evaluate the Immunogenicity, Safety and Optimal Dose of Three Doses Regimen of Recombinant Influenza H5N1 Vaccine, After Two Vaccinations Given 3 Weeks Apart, in Healthy Young Adults.
Brief Title: Immunogenicity, Safety and Optimal Dose Finding Study of Recombinant Influenza H5N1 Vaccine in Healthy Young Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UMN Pharma Inc. (Industry)
Responsible Party: Clinical Development Department, UMN Pharma Inc.
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: JPIP501-01a
Record Dates: First submitted 2009-09-17; First posted 2009-09-21 (Estimated); Last update posted 2010-02-08 (Estimated); Status verified 2010-02

CONDITIONS: Influenza; Virus Diseases
Keywords: H5N1; Vaccine; Influenza H5N1; Avian influenza H5N1; Pandemic
MeSH Terms: conditions — Influenza, Human; Virus Diseases | interventions — FluBlok

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- UMN-0501 45µg (Experimental): Recombinant H5N1 vaccine 45µg
  Interventions: Biological: UMN-0501
- UMN-0501 90µg (Experimental): Recombinant H5N1 vaccine 90µg
  Interventions: Biological: UMN-0501
- UMN-0501 135µg (Experimental): Recombinant H5N1 vaccine 135µg
  Interventions: Biological: UMN-0501

INTERVENTIONS:
Biological: UMN-0501 — 2 doses of recombinant H5N1 A/VN/1203/2004 vaccine 45µg three weeks apart
  Other Names: UMN-05
  Arms: UMN-0501 45µg
Biological: UMN-0501 — 2 doses of recombinant H5N1 A/VN/1203/2004 vaccine 90µg three weeks apart
  Other Names: UMN-05
  Arms: UMN-0501 90µg
Biological: UMN-0501 — 2 doses of recombinant H5N1 A/VN/1203/2004 vaccine 135µg three weeks apart
  Other Names: UMN-05
  Arms: UMN-0501 135µg

SUMMARY:
UMN-0501 is a purified recombinant influenza HA vaccine (A H5N1/Vietnam/1203/2004).

The purpose of the present study is to evaluate immunogenicity, safety and optimal dose among three different doses of UMN-0501 following two same-dose vaccinations of UMN-0501 per patient with a 3 week interval between vaccination in healthy young adults.

Immunogenicity will be confirmed by both microneutralization (MN) antibody and hemagglutination inhibition (HAI) titer levels in the serums of subjects after receiving different doses of UMN-0501. There will be three dose groups with 30 subjects per group for a total of 90 healthy young adults aged 20-40 years enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult as determined by medical history, physical examination, laboratory test, and clinical judgment of the investigator.
* Males and females aged 20-40 years.
* Provides signed informed consent form after received a detailed explanation of the study protocol prior to any study procedures.

Exclusion Criteria:

* Body Mass Index (BMI) 30 kg/m2 and above.
* Has a history of a A/H5N1 influenza virus infection and subjects had received other A/H5N1 influenza vaccine.
* Has a history of allergic reaction by food and medicine including vaccine, and acute fever illness (greater than 39.0C) within 2 days of vaccination.
* Has a history of Guillain-Barre syndrome or acute disseminated encephalomyelitis (ADEM).
* Has severe allergic diseases.
* Has asthma.
* Has a history of convulsions.
* Has a history of any serious disease.
* Known impairment of imune function.
* Known rheumatism and autoimmune disease.
* Receipt of medicines that would affect evaluation of immunogenicity.
* Receipt of any live virus vaccination or receipt of any inactivated vaccine/toxoid prior to enrollment.
* Blood donation prior to enrollment.
* Receipt of another investigation agent prior to enrollment.
* History of alcohol or drug abuse.
* Females who are pregnant or potentially childbearing or are breastfeeding.
* Ineligible subject based on the judgement of the investigator.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2009-10; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Number of subjects who achieve seroconversion, seroprotection, GMTs and GMT ratio to baseline, 21 days after the 2nd vaccination defined by serum neutralizing and HAI titers against the influenza H5N1 A/Vietnam/1203/2004 virus. | Day 42: 21 days after 2nd vaccination (42 days after 1st vaccination)
Frequencies of AEs including vaccine-related reactogenicity events. | Throughout study period: Day0 to 42

SECONDARY OUTCOMES:
To explore T-cell response in the subset of subjects after each vaccination as determined by proliferation and cytokine production capacity of T-cells re-stimulate by H5N1 A/Vietnam/1203/2004 recombinant virus antigens. | Day0, Day 21 and Day 42

CONTACTS AND LOCATIONS:
Overall Officials: Tetsuo Nakayama, MD, PhD, Study Director — Kitasato University Kitasato Institute for Life Sciences; Suminobu Ito, MD, PhD, Principal Investigator — National Hospital Organization
Locations (2):
- Japan (2):
  - National Hospital Organization Osaka Minami Medical Center, Kawachi-Nagano, Osaka
  - National Hospital Organization Tokyo Medical Center, Meguro-ku, Tokyo